CLINICAL TRIAL: NCT02733991
Title: Study of MiniMed™ 640G Insulin Pump With SmartGuard™ in Prevention of Low Glucose Events in Adults With Type 1 Diabetes
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP311
Record Dates: First submitted 2016-03-29; First posted 2016-04-12 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): MiniMed™640G and Suspend before Low feature of SmartGuard™ turned on.
  Interventions: Device: MiniMed™640G and Suspend before low
- Control (Active Comparator): MiniMed™640G alone
  Interventions: Device: MiniMed™640G

INTERVENTIONS:
Device: MiniMed™640G and Suspend before low — All enrolled subjects will start a run in phase, receive training and start pump therapy with the MiniMed™640G insulin pump and usage of blinded Continuous Glucose Monitoring. Eligible subjects that meet the randomization criteria assessed after the running phase will be randomized into the treatment or control arm. Treatment Arm: training and start of Sensor Augmented Pump therapy with Suspend before Low feature of SmartGuard turned ON.
  Control Arm: continuation of pump therapy alone with blinded continuous glucose monitoring for a total of 6 weeks during the treatment phase.
  Other Names: MiniMed™640G and SmartGuard™; MiniMed™640G and Predictive Low Glucose Management
  Arms: Treatment
Device: MiniMed™640G — Control Arm: continuation of pump therapy alone with blinded continuous glucose monitoring for a total of 6 weeks.
  Arms: Control

SUMMARY:
A premarket, international multicenter, prospective, open label, adaptive, randomized controlled study.

The aim is to evaluate the efficacy of sensor augmented pump therapy with MiniMed™640G and SmartGuard™in preventing hypoglycemic events in comparison with continuous subcutaneous insulin infusion therapy in type 1 diabetes adults with an increased risk of hypoglycemia. The primary objective is to demonstrate a reduction in the mean number of hypoglycemic events when using the MiniMed™640G system with SmartGuard™ and the secondary objectives will aim at evaluating the difference in glycemic parameters and HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Age 24-75 years old at time of screening.
* Diagnosed with Type 1 diabetes ≥10 years prior to screening.
* On pump therapy for ≥ 6 months prior to screening.
* Not on Real Time continuous glucose monitoring for ≥ 3 months prior to screening.
* HbA1c value ≥5.8% and ≤10.0% as assessed by local lab ≤ 15 days prior to screening or performed at screening.
* A documented Severe Hypoglycemia event ≤ 12 months prior to screening, OR Clarke score ≥4 assessed at time of screening, OR
* Gold score ≥4 assessed at time of screening.
* Subject is willing to sign and date informed consent, comply with all study procedures and wear all study devices as required during the study.

Exclusion Criteria:

* Untreated Addison's disease, thyroid disorder, growth hormone deficiency, hypopituitarism or definite gastroparesis, per investigator judgment.
* Subject is using Pramlintide (Symlin) SGLT2 inhibitor, GLP agonist at time of screening.
* Renal failure defined by creatinine clearance <30 ml/min, as assessed by local lab test ≤ 3 months before screening or performed at screening at local lab.
* Hearing or vision impairment hindering perception of glucose display and alarms, or otherwise incapable of using the study devices, per investigator judgment.
* Current pregnancy or intention to conceive.
* Any unresolved adverse skin condition in the area of sensor placement (e.g. psoriasis, rash, Staphylococcus infection).
* Alcohol or drug abuse, other than nicotine, per investigator judgment.
* Any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
* Legally incompetent, illiterate or vulnerable person.

Randomization Criteria:

* If subjects meet the above criteria, as well as all of the following criteria assessed at the end of the run-in period, they may continue to participate in the treatment period of the study:

  * Subject has worn two weeks the sensor with transmitter during the run-in period.
  * Subject has shown acceptable tolerance of sensor wear, per investigator judgment.
  * Subject performed ≥ 4 finger stick blood glucose measurements daily, as determined by CareLink™ Clinical data upload as the mean number of SMBG/day over the past 14 days (SMBG number / day ≥ 3.5 rounds up to 4).
  * Subject showed ability to comprehend the pump training and study procedures, per investigator judgment.

Ages: 24 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- France (4):
  - CHU de Besançon, Besançon
  - CHU Grenoble, Grenoble
  - APHM - La Conception, Marseille
  - CHU Montpellier - Hôpital Lapeyronie, Montpellier
- Italy (3):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Ospedale S. Raffaele, Milan
  - Ospedale S. Gionanni di Dio, Olbia
- Netherlands (4):
  - Groene Hart Ziekenhuis, Gouda
  - Maasstad Ziekenhuis, Rotterdam
  - UMC Utrecht, Utrecht
  - Isala, Zwolle
- United Kingdom (3):
  - Harrogate District Hospital, Harrogate, N. Yorkshire
  - King's College London, London
  - Manchester Diabetes Center, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habteab A, Castaneda J, de Valk H, Choudhary P, Bosi E, Lablanche S, de Portu S, Da Silva J, Vorrink-de Groot L, Shin J, Cohen O. Predicting Factors Associated with Hypoglycemia Reduction with Automated Predictive Insulin Suspension in Patients at High Risk of Severe Hypoglycemia: An Analysis from the SMILE Randomized Trial. Diabetes Technol Ther. 2020 Sep;22(9):681-685. doi: 10.1089/dia.2019.0495. PMID 32412858
- [Derived] Bosi E, Choudhary P, de Valk HW, Lablanche S, Castaneda J, de Portu S, Da Silva J, Re R, Vorrink-de Groot L, Shin J, Kaufman FR, Cohen O; SMILE Study Group. Efficacy and safety of suspend-before-low insulin pump technology in hypoglycaemia-prone adults with type 1 diabetes (SMILE): an open-label randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Jun;7(6):462-472. doi: 10.1016/S2213-8587(19)30150-0. Epub 2019 Apr 29. PMID 31047902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 76 | 77
Completed | 75 | 72
Not Completed | 1 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 70 | 135
  >=65 years | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12.22) | 47.4 (12.53) | 48.2 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 38 | 39 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 15 | 15 | 30
  Italy | 19 | 20 | 39
  United Kingdom | 16 | 14 | 30
  France | 14 | 16 | 30
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Sensor Glucose Hypoglycaemic Events Below or Equal to 55 mg/dL Per Patient/Week.
Time Frame: 6 months
Population: 2 participants in the control arm did not have data.
Measure: Mean (Standard Deviation); unit: hypoglycaemic events per week
Arm/Group | Treatment | Control
Number analyzed (Participants) | 76 | 75
hypoglycaemic events per week | 1.12 (1.229) | 4.13 (3.361)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.88, 95% CI 2-sided [-3.51 to -2.25] — Model based Estimated mean; Treatment arm - Control arm

2. Secondary Outcome: Mean Time Spent of Sensor Glucose Values Below or Equal 55 mg/dL.
Time Frame: 6 months
Population: 2 participants in the control arm did not have data.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Treatment | Control
Number analyzed (Participants) | 76 | 75
minutes per day | 12.85 (12.741) | 60.08 (53.644)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -42.62, 95% CI 2-sided [-52.01 to -33.19] — Model based Estimated mean; Treatment arm - Control arm

3. Secondary Outcome: Mean Time Spent of Sensor Glucose Values Within Range and Including 70-180 mg/dL.
Time Frame: 6 months
Population: 2 participants in the control arm did not have data.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Treatment | Control
Number analyzed (Participants) | 76 | 75
minutes per day | 862.91 (162.910) | 832.18 (168.690)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Non-Inferiority — Non-inferiority margin of 40 min/day; Mean Difference (Final Values) = -38.8, 97.5% CI 1-sided [upper limit -0.46] — Model based Estimated mean; difference = control arm - treatment arm
Statistical Analysis 2: Comparison: Treatment vs Control; Test type: Superiority; p = 0.0474, Mixed Models Analysis; Mean Difference (Final Values) = 38.8, 95% CI 2-sided [0.46 to 77.11] — Model based Estimated mean; Difference = Treatment arm - Control arm

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 6/76 | 1/77
Other Adverse Events (participants affected / at risk) | 36/76 | 37/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=76) | Control (N=77)
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anterior cruciate ligament tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=76) | Control (N=77)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Polyuria-polydipsia syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Left cataract (Eye disorders) | 1 (1) | 0 (0)
Eye ulcer (Eye disorders) | 1 (1) | 0 (0)
Swelling abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Antibiotic-associated diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cannula site pain (General disorders) | 0 (0) | 1 (1)
Device intolerance (General disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 0 (0) | 1 (1)
Injection site lump (General disorders) | 1 (1) | 0 (0)
Medical device site erythema (General disorders) | 1 (1) | 1 (1)
Medical device site bleeding (General disorders) | 4 (4) | 3 (3)
Medical device site irritation (General disorders) | 3 (3) | 1 (1)
Medical device site pain (General disorders) | 1 (1) | 2 (2)
Medical device site pruritus (General disorders) | 1 (1) | 2 (2)
Medical device site reaction (General disorders) | 1 (2) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Flu syndrome (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 1 (1)
Common cold (Infections and infestations) | 2 (4) | 3 (4)
Rhinopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Belly button infection (Infections and infestations) | 1 (1) | 0 (0)
Cold sores (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured toe (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured metacarpal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Leg injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (9) | 5 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 10 (18)
Generalised joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fascitis plantar (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Light headedness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intermittent headache (Nervous system disorders) | 0 (0) | 1 (1)
Mood disorder NOS (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Depression worsened (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lipodystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching both hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Medial sclerosis (Vascular disorders) | 1 (1) | 0 (0)
Bleeding (Vascular disorders) | 0 (0) | 1 (1)
Hypertension worsened (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure low (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02733991/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02733991/SAP_001.pdf